CLINICAL TRIAL: NCT00196768
Title: Treatment of Relapsed Acute Promyelocytic Leukemia With Arsenic Trioxide (Phase IV Study)
Brief Title: Treatment Protocol for Relapsed Acute Promyelocytic Leukemia (APL) With Arsenic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: German AML Cooperative Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30052004
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Relapsed Acute Promyelocytic Leukemia; Refractory Acute Promyelocytic Leukemia
Keywords: relapsed; acute promyelocytic leukemia; arsenic
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Recurrence | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic trioxide
Drug: Trisenox

SUMMARY:
Summary

Acute promyelocytic leukemia is defined by a characteristic morphology (AML FAB M3/M3v), by the specific translocation t(15;17) and its molecular correlates (PML/RARa and RARa/PML). Thereby it can be separated from all other forms of acute leukemia.

By all-trans retinoic acid in combination with chemotherapy cure rates of 70 to 80% can be reached. On average, about 10% of patients still die in the early phase of the treatment and about 20 to 30% relapse. Molecular monitoring of the minimal residual disease (MRD) by qualitative nested RT-PCR and quantitative REAL-time PCR of PML/RARa allows to follow the individual kinetics of MRD and to identify patients with an imminent hematological relapse.

A standardized treatment for patients with relapsed APL has not yet been established. With arsenic trioxide (ATO) monotherapy remission rates over 80% were achieved and long-lasting molecular remissions are described. The drug was mostly well tolerated. ATO exerts a dose dependent dual effect on APL blasts, apoptosis in higher and partial differentiation in lower concentrations. ATO was also successfully administered before allogeneic and autologous transplantation. ATO is approved for the treatment of relapsed and refractory APL in Europe and in the USA.

In the present protocol, ATO is given for remission induction:

1. in patients with hematological or molecular first or subsequent relapse of APL and
2. in patients who do not reach a hematological or molecular remission after first line therapy.

Induction therapy with ATO is the mandatory part of the protocol.

After remission induction, there are several options for postremission therapy. Factors which have influence on the treatment decision in the individual case are:

1. the eligibility for allogeneic transplantation
2. the eligibility for autologous transplantation
3. the presence or absence of contraindications against intensive chemotherapy
4. the PCR status after induction and during follow up (RT-PCR of PML/RARa, sensitivity 10-4)

A mandatory form of post-remission therapy is not defined in the protocol. Data and outcomes of any post-remission therapy should be documented in order to collect data of treatment after ATO.

The following stratification of post-remission therapy can be performed according to the decision of the treating physician:

Patients with a HLA-compatible donor who are suitable for allogeneic stem cell transplantation should be transplanted. In patients with a positive PCR one cycle of intensive chemotherapy (HAM) before transplantation should be considered and patients with a negative result are immediately transplanted without preceding chemotherapy. In patients who do not qualify for allogeneic, but for autologous transplantation, the intensity of the chemotherapy (Ara-C dose of the HAM cycle) is scheduled according to the PCR status after ATO and to the patient's age. In patients under 60 years, the recommended single Ara-C dose is scheduled to 3 g/m² in case of a positive PCR result and to 1 g/m² in case of a negative PCR result after ATO. In all patients aged over 60 years, the Ara-C dose should be uniformly reduced to 1 g/m² independent of the PCR status. Patients who are not eligible for allogeneic or autologous transplantation (too old, no stem cells collected, PCR positive stem cell transplant, contraindications against intensive chemotherapy) receive three further cycles with ATO and ATRA. The group of patients not qualifying for autologous transplantation, but without contraindications against intensive chemotherapy should receive an age adapted HAM, whenever a positive PCR persists or reappears after the three maintenance cycles of ATO. A close monitoring of the PCR of PML/RARa after each treatment cycle is part of the protocol.

The main objective of the protocol is to take advantage of the expected low toxicity of ATO and to keep the part of chemotherapy as low as possible.

DETAILED DESCRIPTION:
Synopsis

Title of study

Treatment of acute promyelocytic leukemia (APL) with arsenic trioxide (ATO). A phase-IV study to assess the effectiveness and toxicity of ATO as well as the kinetics of minimal residual disease (MRD) in patients with first and subsequent hematological or molecular relapse of APL.

Study coordination: Priv.-Doz. Dr. Eva Lengfelder

Protocol committee: German AMLCG and German AML-Intergroup (open for other participating groups)

Study duration: Time of recruitment 3 years, individual follow up scheduled for 3 years

Objectives of the study

Primary objectives

Assessment of:

1. the rate of hematological remission
2. the rate of molecular remission
3. the kinetics of the MRD of PML/RARa during and after ATO

Secondary objectives

Assessment of:

1. the side effects of ATO
2. percentage of transplantable patients in comparison to the historical results after chemotherapy
3. the overall survival
4. duration of the hematological and molecular remission

   Study characteristics: Open-label multicenter controlled phase-IV study

   Number of patients: 30 patients

   Inclusion criteria

   * Patients in first or subsequent hematological or molecular relapse of APL

   * Persistence of a positive PCR or no hematological CR after first line therapy

   * No complete hematological remission after first line therapy

   * Age over 18 years

   * No upper age limit

   * Informed consent of the patient

   Exclusion criteria

   * Absolute QTc-interval prolonged over 460 msec before therapy (normal electrolytes, no other drugs prolonging the QT-interval )

   * Heart failure NYHA grade III and IV

   * Renal or hepatic failure WHO grade >= III

   * Pneumonia with hypoxemia

   * Uncontrolled sepsis

   * Pregnancy and lactation period
   * Secondary malignancy, which will have major influence on the prognosis
   * Expected noncompliance
   * No informed consent of the patient

   Diagnostic measures:

   Confirmation of relapse by RT-PCR of PML/RARa and by cytogenetics. Follow up PCRs with quantitative nested RT-PCR and qualitative REAL-time PCR of PML/RARa.

   Treatment plan

   Induction therapy:

   - 3 cycles of ATO with the aim to induce a hematological or a molecular remission.

   Options for postremission therapy:

   · Allogeneic transplantation (PBSCT) in suitable patients with a related or unrelated donor.

   The administration of chemotherapy preceding allogeneic transplantation is stratified according to the PCR status after ATO. Chemotherapy (HAM) should be considered in PCR positive patients according to the individual situation.

   No chemotherapy is given in PCR negative patients.

   · Autologous PBSCT in patients without a donor qualifying for autologous transplantation.

   The intensity of chemotherapy (HAM with either 3 or 1 g/m²) is proposed according to the PCR status of PML/RARa (sensitivity 10-4) after ATO and to patient's age.

   · 3 maintenance cycles of ATO. This is followed by HAM in patients with persistence or reappearance of a positive PCR.

   Patients not eligible for allogeneic or autologous transplantation, but without contraindications against intensive chemotherapy. · 3 maintenance cycles of ATO in patients not eligible for allogeneic or autologous transplantation (no suitable donor, too old, no stem cells collected, positive stem cell transplant) and with contraindications against intensive chemotherapy.

   Monitoring of MRD is mandatory after each ATO cycle and further treatment step. (Details of the treatment plan are shown in the overview of the study design, Paragraph 2.2).

   Criteria for evaluation

   The effectiveness of the therapy is assessed by the evaluation of the rate of hematological and molecular remission and of the duration of remission according to the commonly used definitions.

   The safety of the therapy is assessed by a close study monitoring using the criteria of toxicity according to WHO.

ELIGIBILITY:
Inclusion Criteria:

* Patients in first or subsequent hematological or molecular relapse of APL
* Persistence of a positive PCR or no hematological complete remission (CR) after first line therapy
* No complete hematological remission after first line therapy
* Age over 18 years
* No upper age limit
* Informed consent of the patient

Exclusion Criteria:

* Absolute QTc-interval prolonged over 460 msec before therapy (normal electrolytes, no other drugs prolonging the QT-interval)
* Heart failure New York Health Association grade III and IV
* Renal or hepatic failure World Health Organization grade >= III
* Pneumonia with hypoxemia
* Uncontrolled sepsis
* Pregnancy and lactation period
* Secondary malignancy, which will have major influence on the prognosis
* Expected noncompliance
* No informed consent of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Study Completion 2010-12

PRIMARY OUTCOMES:
the rate of hematological remission
the rate of molecular remission
the kinetics of the MRD of PML/RARa during and after ATO

SECONDARY OUTCOMES:
the side effects of ATO
percentage of transplantable patients in comparison to the historical results after chemotherapy
the overall survival
duration of the hematological and molecular remission

CONTACTS AND LOCATIONS:
Overall Officials: Eva Lengfelder, MD, PhD, Principal Investigator — German AMLCG
Locations (1):
- Eva Lengfelder, MD, PhD, Mannheim, Germany

REFERENCES:
- [Derived] Toft P, Olsen HT, Jorgensen HK, Strom T, Nibro HL, Oxlund J, Wian KA, Ytrebo LM, Kroken BA, Chew M. Non-sedation versus sedation with a daily wake-up trial in critically ill patients receiving mechanical ventilation (NONSEDA Trial): study protocol for a randomised controlled trial. Trials. 2014 Dec 20;15:499. doi: 10.1186/1745-6215-15-499. PMID 25528350